CLINICAL TRIAL: NCT03705858
Title: Postremission Therapy With Actinium-225 (225Ac)-Lintuzumab (Actimab-A®) in Patients With Acute Myeloid Leukemia
Brief Title: Actinium-225-Lintuzumab in Patients With Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to difficulty in finalizing the contract
Sponsor: Joseph Jurcic (Other)
Responsible Party: Sponsor-Investigator, Joseph Jurcic, Assistant Professor of Medicine at the Columbia University Medic, Dept of Med Hematology & Onc, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAR9075
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Actinium-225; Lintuzumab; Columbia; Post-remission; Phase I
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ac-lintuzumab (Experimental): Subjects with AML will receive Ac-lintuzumab.
  Interventions: Drug: Ac-Lintuzumab

INTERVENTIONS:
Drug: Ac-Lintuzumab — 225Ac-lintuzumab will administered at 4 dose levels: 0.25, 0.5, 0.75 or 1 µCi/kg intravenously (IV) over 30 ± 10 minutes. The starting dose will be 0.5 µCi/kg. A dose of 0.25 µCi/kg will be studied only if 0.5 µCi/kg is determined to exceed the MTD. The lintuzumab dose will be adjusted to maintain a specific activity of 0.16 µCi/µg
  Other Names: Actimab-A ®

SUMMARY:
The purpose of this study is to see what dose of 225Ac-lintuzumab is safest to give to acute myeloid leukemia (AML) patients who are in remission but still have minimal residual disease (MRD). About 12 subjects will be asked to take part in this phase 1, 3+3 dose-escalation study. In addition to confirming the safety profile of postremission therapy with 225Ac-lintuzumab, preliminary evidence of efficacy will be assessed by estimating progression-free survival (PFS) and overall survival (OS), and serially evaluating for MRD using cytogenetics, fluorescence in situ hybridization (FISH), or flow cytometric assays, as applicable.

DETAILED DESCRIPTION:
Therapy with α particle-emitting constructs of the anti-CD33 monoclonal antibody lintuzumab has demonstrated significant tumor effects in AML. Because therapy is selectively targeted to leukemic blasts, it has the potential advantage of less extramedullary toxicity than conventional systemic agents. Moreover, the unique radiobiological features of α particle emissions may permit more efficient tumor cell kill with greater specificity than treatment with β particle-emitting radioisotopes. Objective responses in AML following treatment with 225Ac-lintuzumab have been seen in cytoreduced disease, either following chemotherapy or using a fractionated dosing scheme.

The presence of MRD detectable by cytogenetic techniques and flow cytometric assays indicates a high risk of relapse for AML patients, despite achieving a clinical complete remission. The high linear energy and short range of α emissions make them ideally suited to eradicate MRD, as suggested by the clinical responses observed in earlier studies. To date, 225Ac-lintuzumab has only been studied in patients with overt leukemia. The aim of this phase 1 study is to identify the maximum tolerated dose (MTD) of 225Ac-lintuzumab that can be given safely to AML patients in the postremission setting in order to eliminate detectable MRD and ultimately prolong PFS and OS.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologically confirmed AML in first, second, or third clinical CR/CRp after any standard or investigational therapy.
2. Subjects must have detectable MRD by cytogenetics, FISH, or flow cytometry after the completion of all planned therapy. Detectable MRD by flow cytometry is defined by the presence of a myeloid blast population with an atypical immunophenotype, constituting less than 5% of all events. Examples of planned therapy courses include induction chemotherapy with cytarabine and an anthracycline followed by consolidation chemotherapy or 4-6 cycles of a hypomethylating agent-based regimen.
3. At the time of diagnosis or most recent relapse, greater than 25% of bone marrow blasts must have been CD33 positive.
4. Age ≥18 years. Because no dosing or adverse event data are currently available on the use of 225Ac-lintuzumab in patients <18 years of age, children are excluded from this study.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
6. Subjects must have adequate bone marrow and organ function documented within 14 days of study entry as follows:

   1. Absolute neutrophil count (ANC) ≥ 1,000/μL;
   2. Platelet count ≥ 50,000/μL;
   3. Serum creatinine ≤ 1.5 × upper limit of normal (ULN) or estimated glomerular filtration rate of > 50 mL/min;
   4. Serum total bilirubin ≤ 1.5 × ULN (unless attributable to Gilbert's disease);
   5. Alkaline phosphatase, serum aspartate aminotransferase (AST), and serum alanine aminotransferase (ALT) ≤ 2.5 × ULN.
7. The effects of 225Ac-lintuzumab on the developing human fetus are unknown. Since radiation exposure, however, is known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of treatment on study. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of 225Ac-lintuzumab administration.
8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Subjects with acute promyelocytic leukemia or BCR-ABL-positive leukemia.
2. Subjects who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. Prior clofarabine is not allowed due to risk of liver dysfunction.
3. Subjects who have previously received 225Ac-lintuzumab.
4. Subjects with an human leukocyte antigen (HLA)-compatible donor or stem cell source who are immediate candidates for allogeneic hematopoietic cell transplantation (HCT).
5. Subjects who are receiving any other investigational agents concurrently.
6. Subjects with active central nervous system (CNS) involvement by AML.
7. Uncontrolled intercurrent illness including, but not limited to, active serious infections uncontrolled by antibiotics, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, documented liver cirrhosis, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Active malignancy within 3 years of study entry, except previously treated melanoma grade 2 or less, non-melanoma skin cancer, carcinoma in situ or cervical intraepithelial neoplasia, and organ confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) levels and are not on active therapy.
9. Prior organ transplant, including allogeneic HCT.
10. Pregnant or nursing women.
11. Subjects with known human immunodeficiency virus (HIV) infection, active hepatitis B, or active hepatitis C.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of postremission therapy | Up to 2 years
  The 3+3 dose-escalation is designed to establish the MTD of postremission therapy with 225Ac-lintuzumab in patients with AML in first, second, or third CR/CRp who have detectable minimal residual disease (MRD) and have completed all planned therapy.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 3 years
  The length of time during and after the treatment of AML that a subject lives with the disease but it does not get worse. It will be calculated from the time of study entry to relapse, death or last follow-up. That includes subjects with at least one cycle of therapy.
Overall Survival (OS) | Up to 3 years
  The Length of time in days during and after the treatment of AML that a subject lives. It will be calculated from the time of entry onto study to death or last follow-up. That includes all subjects who receive at least one cycle of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Jurcic, MD, Principal Investigator — Columbia University/Herbert Irving Cancer Center

IPD SHARING:
Plan to Share IPD: Undecided